CLINICAL TRIAL: NCT06910982
Title: Chronic Low Back Pain Management: Clinical and Psychophysiological Outcomes of Multimodal Approaches - A Randomized Controlled Trial on Yoga and Mindfulness.
Brief Title: Yoga and Mindfulness for Chronic Low Back Pain: A Randomized Controlled Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Advanced Education & Research Center (Other)
Responsible Party: Principal Investigator, Shamoon Noushad, Lecturer, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CLBP-YM-RCT-2025
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Chronic Low Back Pain; Yoga Therapy; Mindfulness-Based Stress Reduction; Sphinx Pose; Functional Disability

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of four intervention groups:
  * Group A (Sphinx Pose Yoga therapy): Participants will undergo Sphinx Pose Yoga therapy, involving gentle stretching exercises aimed at extending the back and activating muscles along the spine, with sessions occurring thrice weekly.
  * Group B (MBSR): Participants will engage in Mindfulness-Based Stress Reduction (MBSR) sessions, combining mindfulness meditation and stretching to cultivate awareness and reduce stress. Sessions will include mindfulness meditation practices, body scan exercises, gentle yoga movements, and discussions on stress reduction and coping strategies, occurring weekly.
  * Group C (Usual Care): Participants will receive usual care as per The Back Book.
  * Group D (Combined Yoga and MBSR): Participants will receive a combined intervention of Sphinx Pose Yoga therapy and MBSR, incorporating elements from both programs, occurring twice weekly.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sphinx Pose Yoga Therapy (Experimental): participants will undergo Sphinx Pose Yoga therapy involving gentle stretching exercises aimed at extending the back and activating muscles along the spine. Sessions will be conducted three times per week for 12 weeks.
  Interventions: Behavioral: Sphinx Pose Yoga Therapy
- Mindfulness-Based Stress Reduction (MBSR) (Experimental): Participants will engage in weekly MBSR sessions, which include mindfulness meditation, body scan exercises, gentle yoga movements, and stress reduction discussions. The intervention will last 12 weeks.
  Interventions: Behavioral: Sphinx Pose Yoga Therapy
- Usual Care (Active Comparator): Participants will receive usual care as per "The Back Book," which includes standard guidelines for managing chronic low back pain (CLBP) without additional yoga or mindfulness interventions.
  Interventions: Behavioral: Sphinx Pose Yoga Therapy
- Combined Yoga and MBSR (Experimental): Participants will receive a combined intervention consisting of Sphinx Pose Yoga therapy and MBSR, integrating elements from both programs. Sessions will be held twice per week for 12 weeks.
  Interventions: Behavioral: Sphinx Pose Yoga Therapy

INTERVENTIONS:
Behavioral: Sphinx Pose Yoga Therapy — A structured yoga-based intervention focusing on the Sphinx Pose, aimed at improving spinal flexibility and reducing pain. Participants will perform three sessions per week for 12 weeks.

SUMMARY:
Chronic low back pain (CLBP) is a leading cause of disability, significantly impacting quality of life and work productivity. Traditional treatments often provide limited relief, necessitating alternative approaches. This multicenter, parallel-arm, randomized controlled trial (RCT) aims to evaluate the efficacy of Sphinx Pose Yoga Therapy (Yoga), Mindfulness-Based Stress Reduction (MBSR), and their combination in managing CLBP among healthcare providers (HCPs).

Participants will be randomly assigned to one of four groups:

Group A (Yoga Therapy): Sphinx Pose Yoga therapy, practiced three times per week.

Group B (MBSR): Weekly mindfulness meditation, body scan, and gentle stretching.

Group C (Usual Care): Standard treatment guidelines as per The Back Book. Group D (Combined Yoga & MBSR): Integrated approach, practiced twice per week. The study will assess pain intensity, functional disability, quality of life, physiological markers, mental health, and heart rate variability. Outcomes will be measured at baseline (Week 0), post-intervention (Week 12), and follow-up (Week 24). The trial aims to determine whether Yoga, MBSR, or their combination provides superior benefits over usual care in CLBP management.

ELIGIBILITY:
Inclusion Criteria:

* Both genders between 25 to 45 years of age.
* Subjects having low back pain complaints and have visited the healthcare provider in recent days.
* Numerical Pain Rating (NPR) scale score ≥ 2 for their pain intensity.
* Roland Morris Disability Questionnaire subject's score should be ≥ 4.
* Fear Avoidance Beliefs Questionnaire (FABQ) work subscale score must be < 19.

Exclusion Criteria:

* Subjects with high risk for physical injuries during exercise.
* Pregnant and/or lactating females.
* Subjects with musculoskeletal disorders.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline (Week 0), Post-Intervention (Week 12), Follow-up (Week 24).
  Measured using the Numerical Pain Rating (NPR) scale (0-10).
Functional Disability | Baseline (Week 0), Post-Intervention (Week 12), Follow-up (Week 24).
  Assessed via the Oswestry Low Back Pain Disability Questionnaire (0-100%).
Physiological Markers | Baseline (Week 0), Post-Intervention (Week 12), Follow-up (Week 24).
  Cortisol (stress response). β-Endorphins (BE) (pain modulation). Substance-P (SP) (pain neurotransmitter). Interleukin-6 (IL-6) and C-reactive protein (CRP) (inflammation).

SECONDARY OUTCOMES:
Quality of Life (QoL) | Baseline (Week 0), Post-Intervention (Week 12), Follow-up (Week 24).
  Assessed using WHOQOL-BREF
Stress Levels | Baseline (Week 0), Post-Intervention (Week 12), Follow-up (Week 24).
  Measured by Sadaf Stress Scale (SSS) - Physical Stress Subscale.
Depression Symptoms | Baseline (Week 0), Post-Intervention (Week 12), Follow-up (Week 24).
  Evaluated via Beck Depression Inventory (BDI).
Anxiety Levels | Baseline (Week 0), Post-Intervention (Week 12), Follow-up (Week 24).
  Assessed using Generalized Anxiety Disorder 7 (GAD-7) scale.
Heart Rate Variability (HRV) | Baseline (Week 0), Post-Intervention (Week 12), Follow-up (Week 24).
  Measured via wearable biofeedback device.

CONTACTS AND LOCATIONS:
Locations (1):
- Malir University of Science & Technology, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Saleem Y, Noushad S, Ahmed S, Ansari B. Chronic low back pain management: clinical and psychophysiological outcomes of multimodal approaches-a randomised controlled trial on yoga and mindfulness. BMJ Open Sport Exerc Med. 2025 Jun 8;11(2):e002697. doi: 10.1136/bmjsem-2025-002697. eCollection 2025. PMID 40510459